CLINICAL TRIAL: NCT02483455
Title: ALC-919 For The Treatment Of Common Warts (Verruca Vulgaris)
Brief Title: ALC-919 For The Treatment Of Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloce BioPharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-ALC-919-US
Record Dates: First submitted 2015-04-21; First posted 2015-06-29 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Verruca Vulgaris
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALC-919 Topical Solution (Experimental): ALC-919 Topical Solution will be applied twice daily to study area for the treatment of Common Warts
  Interventions: Drug: 2014-ALC-919-US
- Vehicle-Control Topical Solution (Placebo Comparator): Vehicle-Control Topical Solution will be applied twice daily to study area for the treatment of Common Warts
  Interventions: Drug: Vehicle-Control Topical Solution

INTERVENTIONS:
Drug: 2014-ALC-919-US — A topical solution to be applied twice daily for the treatment of Common Warts
  Other Names: ALC-919
  Arms: ALC-919 Topical Solution
Drug: Vehicle-Control Topical Solution — A topical solution to be applied twice daily for the treatment of Common Warts
  Other Names: ALC-Vehicle-Control
  Arms: Vehicle-Control Topical Solution

SUMMARY:
This is a single-center, randomized, double blind, vehicle-controlled phase 2 study of subjects 8 years of age and older with Common Warts (Verruca vulgaris) who desire treatment.

DETAILED DESCRIPTION:
This is a single-center, randomized, double blind, vehicle-controlled phase-2 study of subjects 8 years of age and older with Common Warts (Verruca vulgaris) who desire treatment. A total of four visits are planned including one baseline and three follow-ups. Screening will be done at Visit 1 (Baseline) and all safety and efficacy measurements will be made at all subsequent visits (Visits 2-4).

The primary objective is to evaluate the efficacy of twice daily-applied ALC-919 vs. vehicle in male and female subjects 8 years of age and older with Common Warts (Verruca vulgaris). The primary outcome measure is complete resolution of lesions at the 12 week visit. Secondary outcome measures will include the change in lesion count at the 12 week visit, improvement in the Global Aesthetic Improvement Scale score at the 12 week visit and the safety and tolerability profile of the treatment arm compared to the vehicle arm at each study visit. The safety will be assessed using clinical cutaneous safety exams that will report scaling, dryness and erythema on a scale of 0-3 (0= absent, 1=mild. 2=moderate, 3=severe). Tolerability will be assessed by having subjects answer the treatment tolerability questions at each visit during the treatment period. The tolerability question will be assessed using a 0-3 scale for itching, burning, and stinging.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 8 years or older;
* Individuals with at least 1, but not exceeding 10 Common Wart(s) (Verruca vulgaris) to be treated;
* Individuals whose treatment area is located anywhere on the body except for the following prohibited areas which include: the eye area (including eyelids), lips, mouth cavity, nasal cavity, inner ear, palms of the hands (including periungual area), soles of the feet (including periungual area), or the anogenital area;
* Individuals who are generally in good health as determined by the Principal Investigator;
* Willingness and ability to read, understand, and sign the IRB-approved informed consent form in English after the nature of the study has been fully explained and questions have been answered;
* Individuals who are willing to not start any new products OTC or prescription treatments and discontinue any treatment the Principal Investigator feels may interfere with the evaluation of the test products;
* Individuals who are willing to avoid using cosmetic products, creams, salves, or ointments to the treatment area(s);
* Individuals who are willing and able to thoroughly follow the product use instructions, attend all the scheduled visits and successfully complete the study;
* Individuals who are willing and able to not begin any office based treatments for the duration of the study;
* Individuals who are determined to be free of any systemic or dermatologic disorder, which, in the opinion of the Principal Investigator, will interfere with the study results;
* Female subjects determined to be of child-bearing potential must indicate to the best of their knowledge they are not pregnant and/or lactating nor do they intend to become pregnant during their participation in the study;
* Female subjects with reproductive potential must agree to practice medically acceptable form of birth control during the study;
* A female subject who is post-menopausal (amenorrhea for 12 months prior to the Baseline Visit) is not considered of reproductive potential.

Exclusion Criteria:

* Have warts outside of the treatment area, the eye area (including eyelids), lips, mouth cavity, nasal cavity, inner ear, palms of the hands (including periungual area), soles of the feet (including periungual area), or the anogenital area) or any area that would interfere with study procedures or analyses;
* Have participated in an investigational trial within 30 days prior to enrollment;
* Have received cryotherapy in the treatment area within 30 days prior to enrollment;
* Have required or will require systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days prior to enrollment or during the course of the study. Routine use of inhaled or intranasal corticosteroids during the study is allowed
* Have any uncontrolled current infection;
* Female subject who is pregnant, lactating planning to become pregnant, or is breastfeeding;
* Have any chronic or acute medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk (such as an immunodeficiency or relevant genetic syndrome);
* Have any active malignancy or are undergoing treatment for any malignancy other than non-melanoma skin cancer;
* Individuals who are mentally incompetent, unable or not willing to give written informed consent or meet study requirements;
* Subjects viewed by the Principal Investigator as not being able to complete the study.
* Subjects have a known history of irritation or allergy caused by povidone-iodine
* Have an excessive number of Common Warts (Verruca vulgaris), defined as greater than 10

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Resolution of Common Warts (Verruca vulgaris) in Participants with Twice Daily-Applied ALC-919 vs. Vehicle in Subjects 8 years of Age and Older. | 12 weeks
  The Global Aesthetic Improvement Scale will be used to assess number and appearance of Common Warts at each visit.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability with Twice Daily-Applied ALC-919 vs. Vehicle in Subjects 8 Years of Age and Older with Common Warts (Verruca vulgaris). | 12 weeks
  The Global Aesthetic Improvement Scale will be used to assess number and appearance of Common Warts at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollack, MD, Principal Investigator — Philadelphia Institute of Dermatology
Locations (1):
- Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania, United States